CLINICAL TRIAL: NCT03954639
Title: A Phase 3, Randomized, Double Blinded, Active Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL Admixed With Bupivacaine vs. Bupivacaine Only Administered as Combined Sciatic (in Popliteal Fossa) and Adductor Canal Nerve Block for Postsurgical Analgesia in Subjects Undergoing Lower Extremity Surgeries
Brief Title: Phase 3, Randomized, Double Blinded, Active Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL Admixed With Bupi vs. Bupi Only Administered as Combined Sciatic and Adductor Canal Nerve Block for Postsurgical Analgesia in Lower Extremity Surgeries
Acronym: STRIDE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 402-C-332
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-05

CONDITIONS: Bunion; Metatarsophalangeal Fusion; Midfoot Fusion; Hindfoot Fusion; Total Ankle Arthroplasty; Forefoot Surgery
MeSH Terms: conditions — Bunion | interventions — Suspensions; Injections; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Group 1 (Experimental): Subjects in this group will receive ultrasound guided combined sciatic (in popliteal fossa) and adductor canal nerve block with EXPAREL.
  EXPAREL will be mixed with Bupivacaine
  Subjects enrolled in Cohort 1 will provide blood samples and measures for efficacy and safety.
  Interventions: Drug: EXPAREL 13.3Mg/mL Suspension for Injection
- Cohort 1, Group 2 (Active Comparator): Subjects in this group will receive ultrasound guided combined sciatic (in popliteal fossa) and adductor canal nerve block with bupivacaine.
  Subjects enrolled in Cohort 1 will provide blood samples and measures for efficacy and safety.
  Interventions: Drug: Bupivacaine Hydrochloride
- Cohort 2, Group 1 (Experimental): Subjects in this group will receive ultrasound guided combined sciatic (in popliteal fossa) and adductor canal nerve block with EXPAREL.
  EXPAREL will be mixed with Bupivacaine
  Subjects enrolled in Cohort 2 will provide measures for efficacy and safety.
  Interventions: Drug: EXPAREL 13.3Mg/mL Suspension for Injection
- Cohort 2, Group 2 (Active Comparator): Subjects in this group will receive ultrasound guided combined sciatic (in popliteal fossa) and adductor canal nerve block with bupivacaine.
  Subjects enrolled in Cohort 2 will provide measures for efficacy and safety.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: EXPAREL 13.3Mg/mL Suspension for Injection — Combined Sciatic and Adductor Canal Nerve Block with EXPAREL mixed with Bupivacaine (Single Dose)
  Arms: Cohort 1, Group 1; Cohort 2, Group 1
Drug: Bupivacaine Hydrochloride — Combined Sciatic and Adductor Canal Nerve Block with Bupivacaine HCL
  Arms: Cohort 1, Group 2; Cohort 2, Group 2

SUMMARY:
This is a Phase 3, multicenter, randomized, double blinded, active controlled study in approximately 81 subjects undergoing lower extremity surgeries with combined sciatic and adductor canal nerve block.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages 18 or older
2. American Society of Anesthesiologists (ASA) physical status 1, 2 or 3.
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.
4. Body Mass Index ≥18 and ≤40 kg/m2

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (eg, amide-type local anesthetics, opioids, bupivacaine, NSAIDs)
2. Documented history of long-term diabetes, renal (serum creatinine level >2mg/dL [176.8 μmol/L]) or hepatic dysfunction (serum alanine or aspartame transferase > 3 times the upper limit of normal), coagulation or bleeding disorder and severe peripheral vascular disease
3. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which, in the investigator's opinion may confound the post dosing assessments
4. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
5. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
6. Previous participation in EXPAREL study
7. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance
8. Currently pregnant, nursing, or planning to become pregnant during the study
9. Clinically significant medical disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other conditions that would constitute a contraindication to participation in the study
10. Currently on neuroleptic agent [e.g., gabapentin, pregabalin (Lyrica), duloxetine (Cymbalta) etc.]
11. Inadequate sensory function on the foot (monofilament test)
12. Chronic opioid use in the last 30 days (≥30 morphine equivalents/ day)

    In addition, the subject may be withdrawn from the study if the subject meets the following criterion during or post-surgery:
13. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that, in the opinion of the investigator, renders the subject medically unstable or complicates the subject's post-operative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Magnitude of analgesic effect | 0 hours to 96 hours
  Area under the Curve of the NRS Pain intensity scores from 0 hours to 96 hours post-surgery.

SECONDARY OUTCOMES:
Total Postsurgical Opioid Consumption | 0 hours to 96 hours
  Total Postsurgical opioid consumption from 0 hours to 96 hours post-surgery

IPD SHARING:
Plan to Share IPD: No